CLINICAL TRIAL: NCT05396196
Title: An Analysis of Kinesio® Tape With Manual Fascial Glide Application on Trigger Points in The Iliotibial Band
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Dakota State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IRB0003556
Record Dates: First submitted 2021-06-02; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Myofascial Trigger Point Pain
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pre-Tape (Active Comparator)
  Interventions: Device: Kinesio® Tape
- With Tape 1 (Experimental)
  Interventions: Device: Kinesio® Tape
- With Tape 2 (Experimental)
  Interventions: Device: Kinesio® Tape
- Post-Tape (Experimental)
  Interventions: Device: Kinesio® Tape

INTERVENTIONS:
Device: Kinesio® Tape — Manual Fascial Glide Application

SUMMARY:
Up to 15 participants between the ages of 18-55 will report for two research sessions. Prior to arrival, minimum requirements for being recreationally active or a recreational runner will be confirmed via email using the Pre-Participation Screening form. The first session will require one hour, while the second will require 30 minutes. Maximum amount of time expected is one and a half hours, over two sessions in 48 hours. The 1st and 2nd sessions will be separated by 48 hours. Upon arrival for session 1, informed consent will be obtained along with the following demographic information: age, sex, height, weight, dominant leg, and activity. Participants will then be assessed for trigger points in their dominant side iliotibial band via palpation. Diagnostic criteria for trigger point will be modeled after Travell and Simons: taut band and pain upon palpation. One to four trigger points will be marked on the subject's skin with marker or pen. Pain pressure threshold will be obtained via algometer, using the terminology "Tell me the first moment you experience pain by verbalizing 'now'. Then, three pain pressure threshold readings will be taken per trigger point and then averaged by the researcher. Following, a Visual Analogue Scale for pain will be assessed by asking the question 'On average, on a scale from 0-10 how painful was the pressure?' Kinesiology tape will then be applied to the identified trigger points using the Manual Fascial Glide. The Manual Fascial Glide will be applied with one 'I' strip horizontal to each trigger point. The tape will be anchored adjacent to the marked trigger point, a gentle pressure will be placed on the anchor while applying a lateral glide of the superficial tissue, and adhering the tape in the opposite direction at 30% tension. Pain pressure threshold will be obtained again with the same protocols 10 minutes after the tape is applied. The participant will be asked to wear the tape for 48 hours. Upon arrival for session 2, the application of the tape will be confirmed. Next, a second VAS for pain regarding the previous 48 hours will be completed by the participant. With the participant's choice to continue in the study, a third and fourth measurement of pain pressure threshold will be obtained: one with the tape remaining on, and another 10 minutes after removal of the tape. Again, three pain pressure threshold readings will be taken per trigger point and then averaged by the researcher.

Regarding the new Covid-19 protocols for face-to-face research studies, the following protection guidelines will be followed according to the IRB recommendations. All participants will be seen individually, with no other participants in the research area at the same time. Due to the extended interaction, all participants and researchers will be required to wear a face covering, which covers their mouth and nose at all times while in the research area. The researcher will also wear a face covering over nose and mouth at all times in the research area. This study does not include any high exertion exercise which would increase the risk of infection. Physical distancing of 2 meters between the participant and the researcher will be maintained before and after any necessary close contact evaluation or tape application. All equipment (algometer, computer, examination tables, stools/chairs, pens, scissors, adherent spray bottle, hair trimmer) will be disinfected between each participant. Any disposable equipment (isopropyl alcohol pads, tape, or tape paper) will be disposed of immediately after use. The researcher will wash hands before and after each physical interaction with participants according to the CDC guidelines. Ventilation will be considered in the research area by allowing the door to remain open if the participant allows. Finally, the IRB approved COVID-19 screening questions will be presented to the participant before any part of the research study is completed. If any person answers 'yes' to any of the questions, they cannot participate.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active per the American College of Sports Medicine or Recreational runners will have to report at least 10 miles a week for the last three months.

Exclusion Criteria:

* acute strain or surgery to the knee, quadriceps, or hamstrings
* allergy to adhesive
* malignancies
* cellulitis
* skin infection
* diabetes
* fragile skin

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
with-in subject differences pre- and 10-minute post- tape application measured by pain pressure threshold (N/s2) via algometer | 10 minutes
with-in subject differences pre- and 48-hour post- tape application measured by pain pressure threshold (N/s2) via algometer | 48 hours
with-in subject differences 10-minute post- and 48-hour post- tape application measured by pain pressure threshold (N/s2) via algometer | 48 hours
with-in subject differences 48-hour post- tape application and post- 10- minute tape removal measured by pain pressure threshold (N/s2) via algometer | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- North Dakota State University, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No